CLINICAL TRIAL: NCT03054662
Title: Non Substitutive Strategies to Improve Haemophilia Care in Developing Countries. Experience in Ivory Coast.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: World Federation of Hemophilia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 002/MSHP/CNER-kp
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Haemophilia; Developing Countries
Keywords: Haemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Educational Status; Physical Therapy Modalities; Dental Care; Acetaminophen

STUDY DESIGN:
Intervention Model Description: monocentric prospective study with longitudinal data collection of a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Haemophilia (Experimental): Male patients with severe and moderate haemophilia A and B in Ivory Coast
  Interventions: Other: Education; Diagnostic Test: Improve biological diagnosis and follow-up of haemophilia; Drug: Implement haemostatic non substitutive care of haemophilia; Other: Implement non haemostatic care of haemophilia
- Carriers for Haemophilia (Experimental): Carriers for severe and moderate haemophilia A and B in Ivory Coast
  Interventions: Other: Education; Diagnostic Test: Improve biological diagnosis and follow-up of haemophilia; Drug: Implement haemostatic non substitutive care of haemophilia

INTERVENTIONS:
Other: Education — Education of patients and caregivers about haemophilia and carriers of haemophilia.
Diagnostic Test: Improve biological diagnosis and follow-up of haemophilia — train the laboratory to the diagnosis ans follow-up un haemophilia
Drug: Implement haemostatic non substitutive care of haemophilia — Implement the use of DDAVP and antifibrinolytics in patients with haemophilia and symptomatic carriers
Other: Implement non haemostatic care of haemophilia — Implement regular physiotherapy, develop dental care, promote the regular use of pain killers
  Other Names: Physiotherapy, dental care, pain killers
  Arms: Patients with Haemophilia

SUMMARY:
This study aims to make an inventory of the condition and care of patients with haemophilia and carriers for haemophilia in Ivory Coast and to promote the use non substitutive strategies that are not costly and available in Ivory Coast, to improve the management of haemophilia in this country. The purpose of this project is to evaluate the extent to which the active promotion of these various measures will improve the care of patients with haemophilia and carriers in Ivory Coast.

DETAILED DESCRIPTION:
1. Establish a baseline of the condition of haemophilia in Ivory Coast (number of patients, demographics, reassessment of diagnosis, joint status...).(year 1)
2. Develop tools to assess the intervention (eg transcultural validation of QoL questionnaires, develop booklets to record bleedings...). (year 1)
3. Intervention phase that will focus on education of patients and their family, education of caregivers, training of the laboratory to the diagnosis of haemophilia and promotion of non substitutive strategies to improve haemophilia care in Ivory Coast (DDAVP, antifibrinolytics, physiotherapy, dental care,...).
4. Follow-up phase during 2 years.
5. Outcome analysis

ELIGIBILITY:
Inclusion Criteria:

* Males with severe and moderate haemophilia A and B in Ivory Coast (any age).
* Females over 12 years who are carriers for severe and moderate haemophilia A and B in Ivory Coast.
* Exclusion Criteria: subjects not willing to participate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Improve haemophilia care in Ivory Coast | 2 years after intervention
  Compare QoL questionnaires before and after the intervention phase
Improve haemophilia diagnosis of haemophilia in Ivory Coast | 3 years
  Compare the number of patients with haemophilia between the beginning and the end of the study
Improve haemophilia care in Ivory Coast | 2 years after intervention
  Compare the pain assessment before and after the intervention phase
Improve knowledge about haemophilia in Ivory Coast | 2 years after intervention
  Compare the knowledge queestionnaires about haemophilia before and after the intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Lambert, MD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- CHU de Yopougon, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No